CLINICAL TRIAL: NCT01179269
Title: Pazopanib and Weekly Paclitaxel in Stage IIIB/IV Non-small Cell Lung Cancer
Brief Title: Pazopanib and Paclitaxel for Non-Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped because the research team was unable to enroll any participants
Sponsor: Loyola University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202499
Record Dates: First submitted 2010-08-06; First posted 2010-08-11 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; Pazopanib; Stage IIIB/IV non small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pazopanib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pazopanib plus Paclitaxel (Experimental): Pazopanib daily and weekly Paclitaxel IV.
  Interventions: Drug: Pazopanib plus Paclitaxel

INTERVENTIONS:
Drug: Pazopanib plus Paclitaxel — Pazopanib daily and weekly paclitaxel IV

SUMMARY:
Lung cancer is the leading cause of cancer worldwide with approximately 1.2 million new cases each year. Non-small cell lung cancer (NSCLC) accounts for greater than 80% of all lung carcinomas in Western countries. Surgical resection is the treatment of choice for patients with early stage disease (Stage I and II), but at least 50% of these patients will relapse locally and/or develop distant metastases. Furthermore, 70% of patients with NSCLC are non-resectable at the time of their diagnosis due to either locally advanced or metastatic disease. The long-term prognosis for patients with NSCLC remains poor with the overall 5-year survival rate less than 15%. The low survival rate may be attributed to the high incidence of unresectable disease at presentation and the inability of systemic therapy to cure metastatic disease. There is a clear need for improvement in the treatment of NSCLC.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the objective response rate of pazopanib in combination with paclitaxel in the treatment of subjects with advanced NSCLC. Tumor response will be assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria (version 1.1). A subject is defined as a responder if he/she sustains a complete response (CR) or a partial response (PR) for at least 4 weeks at any time during treatment. A subject without a post-baseline assessment of response will be considered a non-responder.

A secondary objective of this study is to evaluate the safety and tolerability of pazopanib in combination with paclitaxel in the treatment of subjects with advanced NSCLC. Safety and tolerability endpoints will consist of the evaluation of adverse events (AEs), exposure, withdrawals due to AEs, dose reductions or interruptions, and changes from baseline in vital signs and clinical laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of Stage IIIB (with confirmed malignant pleural effusion) or Stage IV NSCLC.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* No prior systemic first-line therapy for Stage IIIB/IV NSCLC with chemotherapy or any other biologic therapy. Prior surgery and/or localized irradiation for NSCLC are permitted. Palliative radiation therapy must have ended 14 days prior to first dose of pazopanib. Subject with recurrence after previous NSCLC that has been treated with surgery with or without adjuvant chemotherapy/radiation for curative intent are eligible, provided 12 months have passed since this treatment ended.

Exclusion Criteria:

* Appropriate for doublet therapy as first line therapy. At discretion of investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Objective response rate of pazopanib in combination with paclitaxel | 2 years
  The count of individuals who sustain a complete response (CR) or a partial response (PR) for at least 4 weeks at any time during two years of treatment will be reported. A CR or PR response will be defined using standard RECIST criteria (version 1.1).

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Shafer, DO, Principal Investigator — Loyola University; Cheryl Czerlanis, MD, Principal Investigator — Loyola University

IPD SHARING:
Plan to Share IPD: No